CLINICAL TRIAL: NCT04520958
Title: Preoperative Psychosocial Support for Postoperative Recovery and Health: Mechanistic Substudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB_00123611
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2019-10

CONDITIONS: Pain, Acute; Pain, Joint; Pain
MeSH Terms: conditions — Acute Pain; Arthralgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness of Breath (Experimental)
  Interventions: Behavioral: Mindfulness of Breath
- Mindfulness of Pain (Experimental)
  Interventions: Behavioral: Mindfulness of Pain
- Cognitive-Behaviorally Based Pain Psychoeducation (Active Comparator)
  Interventions: Behavioral: Cognitive-Behaviorally Based Pain Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness of Breath — Mindfulness of Breath consisted of instruction in focused attention on the breath and metacognitive monitoring and acceptance of discursive thoughts, negative emotions, and pain.
  Arms: Mindfulness of Breath
Behavioral: Mindfulness of Pain — Mindfulness of Pain consisted of instruction in how to (1) zoom in to deconstruct pain into its constituent physical sensations and precisely map each sensation's spatial location, (2) use mindful breathing to zoom out and broaden the field of attention to include previously neglected sensory elements (i.e., spaces within the body that were absent of sensation and pleasant sensations), and (3) shift attention from unpleasant sensations to neutral/pleasant sensations or experiences.
  Arms: Mindfulness of Pain
Behavioral: Cognitive-Behaviorally Based Pain Psychoeducation — Cognitive-Behaviorally Based Pain Psychoeducation consisted of psychoeducation about the link between thoughts, emotions, and behavior and provided instruction in the use logic to dispute maladaptive thoughts about pain that might otherwise exacerbate pain and distress.
  Arms: Cognitive-Behaviorally Based Pain Psychoeducation

SUMMARY:
This was a single site, three-arm, parallel group randomized clinical trial that compared the effect of three preoperative psychosocial interventions on knee and hip replacement patients' preoperative pain intensity and postoperative pain intensity, pain unpleasantness, and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking males or females.
* 18 years old or older
* Patients within the University of Utah Hospital system
* Patients attending Joint Academy to prepare for either hip or knee replacement surgery

Exclusion Criteria:

* Altered mental status due to delirium, psychosis, or pharmacological sedation as determined by clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Preoperative Pain Intensity | Completed immediately before the preoperative intervention and immediately after the preoperative intervention (i.e., 20 minutes)
  Single-item Numeric Rating Scale (0-10), with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Postoperative Pain Intensity | Completed on the evenings of the 2nd, 3rd, 7th, 14th, 21st, and 28th postoperative days.
  Single-item Numeric Rating Scale (0-10), with 0 indicating no pain and 10 representing the most intense pain imaginable.

SECONDARY OUTCOMES:
Change in Postoperative Pain Unpleasantness | Completed on the evenings of the 2nd, 3rd, 7th, 14th, 21st, and 28th postoperative days.
  Single-item Numeric Rating Scale (0-10), with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.
Change in Postoperative Opioid Use | Completed on the evenings of the 2nd, 3rd, 7th, 14th, 21st, and 28th postoperative days.
  Single-item, dichotomously scored (no vs. yes): "Did you take opioid medications in the last 24 hours?"

OTHER OUTCOMES:
Change in Self-Transcendent State | Completed immediately before the preoperative intervention and immediately after the preoperative intervention (i.e., 20 minutes)
  Self-transcendent state was measured with the Nondual Awareness Dimensional Assessment (NADAs; Hanley, Nakamura, & Garland, 2018). The NADAs is a 3-item, Likert type (0-10) self-report scale specifically designed to measure alterations in the experience of self occasioned by mindfulness practice.
Patient Confidence | Completed immediately after the preoperative intervention
  Patients' confidence ("How confident are you that you could effectively use this pain management technique?") in using the pain management technique was assessed with a single item rated on a numeric rating scale (0-10), with 0 indicating no confidence and 10 representing complete confidence.
Patient Intent | Completed immediately after the preoperative intervention
  Patients' intent to use the technique ("How likely are you to use this pain management technique?") to use the pain management technique was assessed with a single item rated on a numeric rating scale (0-10), with 0 indicating no intent and 10 representing absolute intent.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanley AW, Gililland J, Garland EL. To be mindful of the breath or pain: Comparing two brief preoperative mindfulness techniques for total joint arthroplasty patients. J Consult Clin Psychol. 2021 Jul;89(7):590-600. doi: 10.1037/ccp0000657. Epub 2021 Jun 24. PMID 34165999